CLINICAL TRIAL: NCT01515072
Title: Remote Ischemic Preconditioning in Neurological Death Organ Donors
Acronym: RIPNOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Baburao Koneru, MD, MPH, Professor, New Jersey Medical School, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120110125
Record Dates: First submitted 2011-10-28; First posted 2012-01-23 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Organ Transplantation
Keywords: Remote Ischemic Preconditioning; Brain death organ donors; Delayed graft function; Donor management; Pulsatile perfusion
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Remote Ischemic Preconditioning (No Intervention): The donors assigned to this group will receive standard of care of management of brain death donors in each organ procurement organization.
- Remote Ischemic Preconditioning (Experimental): The donors assigned to this group would receive two RIPC interventions. The first one would occur immediately after brain death declaration and consent for organ donation. The second one would occur immediately before commencement of organ recovery. At each occasion RIPC would be induced by 4 cycles of mid-thigh inflation of tourniquet for 5 min followed by deflation for 5 minutes.
  Interventions: Other: RIPC (Remote Ischemic Preconditioning)

INTERVENTIONS:
Other: RIPC (Remote Ischemic Preconditioning) — Remote Ischemic Preconditioning (RIPC) by Inflation of Pneumatic Tourniquet. The intervention will consist of tourniquet inflation on the mid-thigh for 5 minutes, followed by a deflation period of 5 minutes for a total of 4 cycles. The intervention will take place at two time points: First, after determination of brain death and consent for organ donation and again upon incision for organ recovery. The second intervention will occur in a manner identical to the first intervention but in the opposite limb.
  Arms: Remote Ischemic Preconditioning

SUMMARY:
The purpose of this study is to determine whether application of lower limb remote ischemic preconditioning (RIPC) after determination of brain death improves donor stability, organ quality, organ yield, and early post transplant clinical outcomes.

Neurological death donors will be stratified into standard and extended criteria donors (SCD/ECD) and randomized in a 1:1 fashion to RIPC or No intervention. The primary outcome is the number of organs recovered per donor. Secondary outcomes include donor hemodynamic state, donor organ-specific function parameters, pulsatile perfusion parameters, number of organs transplanted per donor, recipient hospital free survival and delayed graft function of kidneys. The sample size is powered to detect a difference of 0.44 organs recovered.

DETAILED DESCRIPTION:
Study Design and Participants The RIPNOD trial was conducted from July 2011 to July 2014 as a prospective randomized trial in two OPOs (in New Jersey and in Texas) in the U.S. The funding organization, institutional review boards and the physician committees of the two organ procurement organizations (OPOs) approved the study. Exemptions for consent from potential recipients and for a data and safety monitoring board were granted. Consent for research was obtained from the donor's next of kin by OPO staff unless a 'first-person' consent existed. The study population consisted of neurological death organ donors. Eligible donors were age > 6 years, in whom death declaration was either imminent or completed, and organ recovery was not expected within 6 hours of enrollment. Donors with severe trauma to lower extremity or on sulfonylurea agents were excluded (Trial Protocol in Supplement).

Procedures Randomization (1:1) to No RIPC or RIPC groups in standard and extended criteria donors (SCD and ECD) strata occurred based on a computer-generated random table of numbers. In Texas, field coordinators performed the randomization through a website and administered the intervention. In New Jersey, research staff performed all trial activities and randomized using opaque, sealed envelopes. Organ recovery teams were informed of the study and sometimes knew of the group assignment. The recipient care teams and recipients were not aware of the group assignment.

The intervention consisted of four cycles of inflation of a tourniquet around mid-thigh to 250 mm Hg for 5 minutes followed by 5 minutes of deflation. The initial intervention occurred in the right thigh as early as possible after declaration of death. The second intervention occurred in the left thigh 24 hours after the initial intervention, or immediately before recovery, if this was earlier. Videoconferences between the two sites helped standardize the intervention before the trial commenced. All decisions regarding donor management, organ recovery, machine perfusion of kidneys, transplantation of organs and care after transplantation were independent of the research teams.

Outcomes and Data Collection The primary outcome was the total number of organs recovered per donor. Secondary outcomes were number of organs transplanted per donor, and changes from baseline to terminal (before aortic cross clamp) in vasopressor support, serum lactate, creatinine clearance, left ventricular ejection fraction, serum troponins, partial pressure of arterial oxygen: fraction inspired oxygen (P:F) ratio, dynamic and static lung compliance, and perfusate flow and resistance in machine perfused kidneys, delayed graft function (DGF) in transplanted kidneys and six-month hospital free survival in all recipients. A score quantified vasopressor support.14 All laboratory tests were performed at donor hospitals. Cockcroft-Gault equation was used to calculate creatinine clearance.15 Donor hospital cardiologists estimated the ventricular ejection fraction in transthoracic echocardiograms. OPO policies dictated machine perfusion of kidneys; perfusion, occurred at a central location in each OPO. Delayed graft function was defined as dialysis in the first week after transplant. Six month hospital-free survival was defined as the number of days recipients survived following the initial discharge after the transplant. All donor data were obtained prospectively from OPO records. Data after transplantation were obtained from the Scientific Registry of Transplant Recipients (SRTR). The SRTR data system includes data on all donors, waitlist candidates, and transplant recipients in the United States, submitted by members of the Organ Procurement and Transplantation Network (OPTN). The Health Resources and Services Administration (HRSA), U.S. Department of Health and Human Services provides oversight to the activities of the OPTN and SRTR contractors.

Sample Size A sample size of 150 donors in each arm was estimated to provide 80% power to detect a difference of 0.44 of an organ recovered and 0.48 of an organ transplanted per donor. The difference criterion was chosen based on published results achieved with hormonal resuscitation in organ donors. 6 Pooled standard deviations (organs recovered: 1.35; organs transplanted: 1.5) from data of two OPOs were used.

Statistical Analyses Intention to treat principle was used in all analyses. Discrete descriptive data are reported as counts and percent and continuous data as means (sd) or medians (interquartile range). Continuous variables were compared using either t, or equivalent non-parametric tests. Categorical variables were compared using chi square tests. Multivariate modeling with backward elimination - linear ones to model RIPC on recovery and transplantation of all (0-8) and abdominal organs (0-5) per donor, and logistic ones to model recovery/transplantation of > 1 thoracic organ per donor and DGF - was performed. Because only seven fewer thoracic organs were transplanted than recovered the model for organs transplanted was used to analyze both outcomes. Donor characteristics of age, sex, race, cause of death, BMI, comorbidities (hypertension, diabetes, alcohol use, and hepatitis C), treatments (insulin, diuretics and steroids) and laboratory parameters (serum creatinine and P:F ratio) and OPO site were predictor variables in organ yield models. Donor age or stratum, cold ischemia, number of human leukocyte antigen mismatches and recipients' characteristics of age, sex, race, BMI, diabetes, hypertension, etiology of renal failure, panel reactive antibody and OPO site were predictor variables in models of DGF. For linear regression models, adjusted R2 was computed and residuals were assessed for normality; the C statistic was used to assess goodness of the fit for logistic regression. Statistical significance was set at p<0.05.

Post Hoc Analyses Rates of acute rejection of kidney during the first six months were compared between the two groups using chi square tests. Kaplan-Meier estimates and log rank tests were used to compare unadjusted outcomes of graft and patient survival at 6, 12 and 24 months. In heart, lung and liver recipients, retransplantation or death was defined as graft loss. In all other organs graft loss was death-censored. Cox proportional hazards models were used to estimate the effect of RIPC on the adjusted hazard ratio for six-month graft loss after controlling for OPO site, donor age or stratum and sex, cold ischemia time, number of antigen mismatches, organ transplanted, and recipient age, sex, race, BMI, diabetes and hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Neurological death donors in whom brain death determination is imminent
2. First person consent or next of kin consent for research
3. Donors >=6 years of age
4. Organ recovery not expected within 6 hours of consent.
5. Both sexes and ethnicities.

Exclusion Criteria:

1. Donation after cardiac death donors (DCD)
2. Live organ donors
3. No first person consent and next of kin decline research consent
4. Donor Age < 6 years
5. Lower extremity trauma or recent amputation
6. Tissue only donors

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baburao Koneru, MD, Principal Investigator — University of Medicine and Dentistry New Jersey-Newark; William K Washburn, MD, Principal Investigator — University of Texas Health Sciences at San Antonio
Locations (2):
- United States (2):
  - Rutgers, The State University of New Jersey, Newark, New Jersey
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The RIPNOD trial was conducted from July 2011 to July 2014 in two organ procurement organizations (OPO) in the U.S. Consent for research was obtained from donors next of kin by the OPO staff unless a 'first person' consent existed.
Groups:
- No RIPC: The donors assigned to this group will receive standard of care of management of brain death donors in each organ procurement organization.
- RIPC: The donors assigned to this group would receive two RIPC interventions. The first one would occur immediately after brain death declaration and consent for organ donation. The second one would occur immediately before commencement of organ recovery. At each occasion RIPC would be induced by 4 cycles of mid-thigh inflation of tourniquet for 5 min followed by deflation for 5 minutes.
  RIPC (Remote Ischemic Preconditioning): Remote Ischemic Preconditioning (RIPC) by Inflation of Pneumatic Tourniquet. The intervention will consist of tourniquet inflation on the mid-thigh for 5 minutes, followed by a deflation period of 5 minutes for a total of 4 cycles. The intervention will take place at two time points: First, after determination of brain death and consent for organ donation and again upon incision for organ recovery. The second intervention will occur in a manner identical to the first intervention but in the opposite limb.
Period: Overall Study
Arm/Group | No RIPC | RIPC
Started | 166 | 155
Completed | 166 (There were 566 total organs transplanted and 248 kidneys transplanted in the No RIPC group.) | 155 (There were 513 total organs transplanted and 235 kidneys transplanted in the RIPC group)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All donors enrolled in both groups were included in the in-between group comparisons of baseline characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | No RIPC | RIPC | Total
Number analyzed (Participants) | 166 | 155 | 321
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44 [29 to 54] | 42 [29 to 51] | 43 [29 to 52]
Age, Customized [Number; unit: participants]
  11-25 | 24 | 34 | 58
  26-35 | 39 | 27 | 66
  36-45 | 26 | 34 | 60
  46-75 | 77 | 60 | 137
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 62 | 121
  Male | 107 | 93 | 200
Race/Ethnicity, Customized [Number; unit: participants]
  White | 97 | 74 | 171
  African-American | 35 | 42 | 77
  Hispanic | 30 | 38 | 68
  Other | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 166 | 155 | 321
Body Mass Index (BMI) [Number; unit: participants] — 2 Categories < 30.0
  =/> 30.0
  participants
    BMI < 30.0 | 126 | 104 | 230
    BMI =/> 30.0 | 40 | 51 | 91
Hepatitis C Antibody [Number; unit: participants] — Serological test for Hepatitis C antibody:
  Yes or No
  participants
    Yes | 7 | 16 | 23
    No | 159 | 139 | 298
Co-Morbidities [Number; unit: participants] — Hypertension: Yes or No
  participants
    Hypertension: Yes | 58 | 48 | 106
    Hypertension: No | 108 | 107 | 215
Central Line Use [Number; unit: participants] — Donors who had Central line in place: Yes or No
  participants
    Yes | 121 | 116 | 237
    No | 45 | 39 | 84
Co-Morbidities [Number; unit: participants] — Diabetes: Yes or No
  participants
    Diabetes: Yes | 19 | 21 | 40
    Diabetes: No | 147 | 134 | 281
Co-Morbidities [Number; unit: participants] — Past or Current Smoker: Yes or No
  participants
    Past or Current Smoker:Yes | 89 | 99 | 188
    Past or Current Smoker:No | 77 | 56 | 133
Steroids Administered [Number; unit: participants] — Steroids Administered: Yes or No
  participants
    Steroids Administered: Yes | 125 | 122 | 247
    Steroids Administered: No | 41 | 33 | 74
Insulin Infusion [Number; unit: participants] — Insulin Infusion: Yes or No
  participants
    Insulin Infusion: Yes | 47 | 42 | 89
    Insulin Infusion: No | 119 | 113 | 232
Declaration of Death to Initial Intervention, Hours [Median (Inter-Quartile Range); unit: hours] — Interval from declaration of brain death to the initial intervention.
  hours | 5.8 [4.2 to 8.8] | 7.3 [5.0 to 12.1] | 6.5 [4.7 to 10.4]
Initial Intervention to Cross Clamp [Number; unit: participants] — 3 Groups:
  1. 5.9-24.0 hours
  2. 24.1-39.5 hours
  3. Data Not Available
  participants
    Intervention to Cross Clamp: 5.9-24.0 hours | 123 | 115 | 238
    Intervention to Cross Clamp: 24.1-39.5 hours | 35 | 25 | 60
    Intervention to Cross Clamp: Data not available | 8 | 15 | 23
Vasopressor Score [Median (Inter-Quartile Range); unit: units on a scale] — A numerical score calculated for number and dose of Vasopressors in use. The score is calculated using the following formula (from Zuppa AF et. al.CRIT CARE MED 2004 Vol. 32 p 2318-2322):
  Vasopressor Score= (dopamine dose[y=ug/kg/min x 1]) + (dobutamine dose [ug/kg/min] x 1) + (epinephrine dose [ug/kg/min] x100) + (norepinephrine dose [ug/kg/min] x 100) + (phenylephrine dose [ug/kg/min] x 100).
  The range for our study was 0-4900 with higher doses indicating higher vasopressor use in the donor.
  Data missing per group:
  No RIPC=2 RIPC=2 Population: Data missing for 2 participants in each arm of the study.
  units on a scale
    number analyzed (Participants) | 164 | 153 | 317
    (all) | 100 [0 to 925.0] | 16.0 [0 to 600] | 37 [0 to 800]
P:F ratio [Median (Inter-Quartile Range); unit: ratio] — P:F ratio: Ratio of partial pressure of arterial oxygen: fraction of inspired oxygen.
  Missing data:
  No RIPC=2 RIPC=4
  ratio | 249.8 [154.8 to 393.0] | 244.0 [152.0 to 387.5] | 248 [154.3 to 389.3]
Ventricular Ejection Fraction [Median (Inter-Quartile Range); unit: proportion ejection fraction] — Ventricular Ejection Fraction
  Missing data:
  No RIPC: 39 RIPC: 31
  proportion ejection fraction | 0.6 [0.55 to 0.65] | 0.59 [0.49 to 0.65] | 0.6 [0.52 to 0.65]
Serum Chemistry: Creatinine [Median (Inter-Quartile Range); unit: mg/dL] — Serum Chemistry: Creatinine, mg/dL
  Missing data:
  No RIPC=3 RIPC=2
  mg/dL | 1.0 [0.7 to 1.6] | 1.1 [0.8 to 1.4] | 1.06 [0.8 to 1.4]
Serum Chemistry: Lactate [Median (Inter-Quartile Range); unit: mg/dL] — Serum Chemistry: Lactate, mg/dL
  Missing data:
  No RIPC= 31 RIPC= 21
  mg/dL | 1.5 [1.1 to 2.4] | 1.6 [1.1 to 2.4] | 1.6 [1.1 to 2.4]
Serum Chemistry: Troponin I [Median (Inter-Quartile Range); unit: ng/ml] — Serum Chemistry: Troponin I, ng/ml
  Missing data:
  No RIPC= 37 RIPC= 29
  ng/ml | 0.28 [0.04 to 1.07] | 0.31 [0.07 to 1.25] | 0.29 [0.05 to 1.18]

OUTCOME MEASURES:

1. Primary Outcome: Number of Organs Recovered Per Donor
Description: Number of organs recovered per organ donor
Time Frame: At time of organ recovery, up to 1 day
Population: Subjects were organ donors enrolled in this multicenter study
Measure: Mean (Standard Deviation); unit: organs recovered per donor
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 166 | 155
organs recovered per donor | 3.79 (1.73) | 3.60 (1.84)
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Sample Size and Power estimation: A sample size of at least 150 donors in each arm was estimated to provide 80% power to detect a difference of 0.44 of an organ recovered and 0.48 of an organ transplanted per donor. The difference criterion was chosen based on published results achieved with hormonal resuscitation in organ donors. 6 Pooled standard deviations (organs recovered: 1.35; organs transplanted: 1.5) from data of two OPOs were used; Test type: Superiority or Other; p = 0.38, t-test, 2 sided — This is an unadjusted comparison. P value < 0.05; Adjusted analyses for the RIPC effect are provided below; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.37 to 0.21] — 0.08 less organs per donor in the RIPC group

2. Secondary Outcome: Number of Organs Transplanted Per Donor
Description: Number of organs transplanted from each organ donor
Time Frame: Within 24 hours of organ recovery
Population: Subjects were organ donors enrolled in this multicenter study
Measure: Mean (Standard Deviation); unit: Organs transplanted from each donor
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 166 | 155
Organs transplanted from each donor | 3.41 (1.90) | 3.31 (1.94)
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Sample Size A sample size of at least 150 donors in each arm was estimated to provide 80% power to detect a difference of 0.44 of an organ recovered and 0.48 of an organ transplanted per donor. The difference criterion was chosen based on published results achieved with hormonal resuscitation in organ donors. 6 Pooled standard deviations (organs recovered: 1.35; organs transplanted: 1.5) from data of two OPOs were used; Test type: Superiority or Other; p = 0.70, t-test, 2 sided — This is an unadjusted analysis. P < 0.05; Adjusted analyses are provided below; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.33 to 0.26] — 0.03 less organs per donor in the RIPC group

3. Secondary Outcome: Change in Vasopressor Score
Description: Changes in the following: Vasopressor usage, serum Lactate, Creatinine clearance, arterial oxygen pressure:fraction of inspired oxygen (P:F) ratios, Lung Compliance, Cardiac biomarkers, ejection fraction (EF) from 2-dimensional Echocardiogram.
  Here we will present data for the change in vasopressor use evaluated using a vasopressor score.
  A numerical score calculated for number and dose of Vasopressors in use. The score is calculated using the following formula (from Zuppa AF et. al.CRIT CARE MED 2004 Vol. 32 p 2318-2322):
  Vasopressor Score= (dopamine dose[y=ug/kg/min x 1]) + (dobutamine dose [ug/kg/min] x 1) + (epinephrine dose [ug/kg/min] x100) + (norepinephrine dose [ug/kg/min] x 100) + (phenylephrine dose [ug/kg/min] x 100).
  The range for our study was 0-4900 with higher doses indicating higher vasopressor use in the donor.
Time Frame: Vasopressor score was determined before aortic cross clamp minus the value prior to the first intervention, an average of 19 hours
Population: Donors in whom vasopressor agent and dose were described in the OPO records before intervention and prior to aortic cross clamp.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 158 | 141
units on a scale | -15.60 [-600 to 0] | -6.00 [-400 to 0]
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney) — P<0.05; This is an unadjusted comparison

4. Secondary Outcome: Change in Serum Lactate
Description: Change in serum lactate levels (mg/dL) from before intervention to the final value
Time Frame: Subjects will be followed from admission to explantation, an average of 4.5 days
Population: Donors in whom at least two serum lactate levels (one before and one after the initial intervention) were available
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 127 | 126
mg/dL | 0.12 [-40 to 0.70] | 0.20 [-40 to 0.60]
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.86, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Creatinine Clearance
Description: Change in creatinine clearance (mL/min by Cockcroft-Gault method) from before intervention to terminal value
Time Frame: Subjects will be followed from admission to explantation, an average of 4.5 days
Population: Donors in whom two serum creatinine values (one before intervention and another after the initial intervention) are available.
Measure: Median (Inter-Quartile Range); unit: mL/min
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 155 | 145
mL/min | 0 [-8.1 to 9.8] | 0 [-10.6 to 14.4]
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney) — P<0.05; This is an unadjusted comparison

6. Secondary Outcome: Change in P:F Ratio
Description: Change in ratio of arterial oxygen pressure:fraction inspired oxygen ratio from before intervention to terminal value
Time Frame: Subjects will be followed from admission to explantation, an average of 4.5 days
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- No RIPC: The donors assigned to this group will receive standard of care of management of brain death donors in each organ procurement organization.
  Any discrepancy in the number of participants is attributed to missing data for some participants
- RIPC: The donors assigned to this group would receive two RIPC interventions. The first occurs immediately after brain death declaration and consent for organ donation. The second one immediately before of organ recovery. At each occasion RIPC would be induced by 4 cycles of mid-thigh inflation of tourniquet for 5 min followed by deflation for 5 minutes.
  RIPC (Remote Ischemic Preconditioning): Remote Ischemic Preconditioning (RIPC) by Inflation of Pneumatic Tourniquet. The intervention will consist of tourniquet inflation on the mid-thigh 5 minutes, followed by a deflation period of 5 minutes for a total of 4 cycles. The intervention occurs at two time points: First, after determination of brain death and consent for organ donation and again upon incision for organ recovery. The second intervention will occur in a manner identical to the first intervention but in the opposite limb.
  Any discrepancy in the number of participants is attributed to missing data for some participants
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 152 | 142
ratio | 6.5 [-57.3 to 86.5] | 0.05 [-74.3 to 96.2]
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney) — P<0.05; This is an unadjusted comparison

7. Secondary Outcome: Change in Dynamic Compliance
Description: Change in dynamic compliance of the lung from before intervention to terminal value
  Cdyn = Dynamic compliance; Vt = tidal volume; PIP = Peak inspiratory pressure (the maximum pressure during inspiration); PEEP = Positive End Expiratory Pressure:
  Cdyn= Vt/PIP - PEEP
Time Frame: Subjects will be followed from admission to explantation, an average of 4.5 days
Measure: Median (Inter-Quartile Range); unit: L/cm H20
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 123 | 123
L/cm H20 | 2.30 [-2.0 to 7.6] | 1.20 [-1.8 to 8.1]
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney) — P<0.05; This is an unadjusted comparison

8. Secondary Outcome: Change in Troponins
Description: Change in serum troponin I (ng/mL) from before intervention to terminal value
Time Frame: Subjects will be followed from admission to explantation, an average of 4.5 days
Population: Only donors in whom two troponin I values (one before intervention and another after the initial intervention) were available were included in this analysis
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 122 | 119
ng/mL | -0.04 [-0.38 to 0] | -0.09 [-0.69 to -0.01]
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney) — P<0.05; This is an unadjusted comparison

9. Secondary Outcome: Pulsatile Perfusion Flow
Description: Perfusate flow (mL/min) in machine perfused kidneys.
Time Frame: Up to 24 hours of machine perfusion
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- No RIPC: Kidneys in this group were recovered from donors in the No RIPC arm. Decisions regarding which kidneys were not and were pumped were made by the OPO.
  Any discrepancy in the number of participants is attributed to missing data for some subjects.
- RIPC: Kidneys in this group were recovered from donors in the RIPC arm. Decisions regarding which kidneys were not and were pumped were made by the OPO.
  Any discrepancy in the number of participants is attributed to missing data for some subjects.
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 49 | 32
mL/min
  Flow at 1 hour, mL/min | 98.58 (32.41) | 89.42 (38.31)
  4 hours | 105.28 (23.75) | 104.03 (40.66)
  8 hours | 117.98 (28.86) | 94.21 (32.64)
  12 hours | 115.19 (20.07) | 106.36 (32.55)
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.53, Regression, Linear — P<0.05; Final flow was modeled on RIPC and adjusted for donor stratum and duration of perfusion; Median Difference (Final Values) = -4.7, 95% CI 2-sided [-10.1 to 19.5] — Data shown above is the the adjusted mean difference in final flow in RIPC group

10. Secondary Outcome: Six Month Hospital Free Survival of All Organ Recipients
Description: Six month hospital-free survival was defined as the number of days recipients survived following the initial discharge after the transplant.
Time Frame: 6 months post-transplant
Population: Recipients of all organs from donors enrolled in the two arms
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 482 | 456
days | 172 [165 to 174] | 171 [165 to 174]
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.97, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Delayed Graft Function (DGF) of Kidney Recipients.
Description: DGF is defined as the need for dialysis within the first week post transplantation.
Time Frame: 7 days post-transplant
Population: Kidney recipients of donors in each arm.
Measure: Number; unit: participants
Units Other Than Participants: Kidney Recipients
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 166 | 155
Number analyzed (Kidney Recipients) | 247 | 235
participants
  DGF: Yes | 45 | 51
  DGF: No | 202 | 184
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.07, Chi-squared — Adjusted analysis with recipient age as a continuous variable, sex, race as black versus not black, body mass index, diabetes, hypertension,antigen mismatches, donor age as a continuous variable and trial site; Odds Ratio (OR) = 1.62, 95% CI 2-sided [0.95 to 2.76]
Statistical Analysis 2: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.36, Chi-squared — Unadjusted analysis

12. Secondary Outcome: Pulsatile Perfusion Parameters
Description: Perfusate resistance (mm Hg/mL/min) in machine perfused kidneys.
Time Frame: Up to 24 hours of machine perfusion
Measure: Mean (Standard Deviation); unit: Resistance, mm Hg/mL/min
Arm/Group | No Remote Ischemic Preconditioning | Remote Ischemic Preconditioning
Number analyzed (Participants) | 49 | 32
Resistance, mm Hg/mL/min
  Resistance at 1 hour, mL/min | 0.29 (0.12) | 0.38 (0.30)
  Resistance at 4 hours, mL/min | 0.25 (0.10) | 0.31 (0.23)
  Resistance at 8 hours, mL/min | 0.22 (0.09) | 0.33 (0.23)
  Resistance at 12 hours, mL/min | 0.22 (0.08) | 0.29 (0.22)
Statistical Analysis 1: Comparison: No Remote Ischemic Preconditioning vs Remote Ischemic Preconditioning; Test type: Superiority or Other; p = 0.006, Regression, Linear; Final resistance was modeled on RIPC and adjusted for donor stratum and duration of perfusion; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [0.03 to 0.17] — Data shown above is the adjusted mean difference in final resistance in the RIPC group

13. Post Hoc Outcome: Acute Kidney Rejection
Description: Diagnosis of rejection as documented in the recipient records in the Scientific Registry of Transplant Recipients (SRTR).
Time Frame: 6 months after kidney transplantation
Population: This outcome was examined in recipients of in SRTR that received kidneys from donors in the RIPNOD trial
Measure: Number; unit: participants
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 247 | 235
participants
  Rejection: Yes | 17 | 13
  Rejection: No | 230 | 222
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.50, Fisher Exact; This is an unadjusted comparison

14. Post Hoc Outcome: Graft Survival
Description: Kaplan-Meier estimates of 6, 12 and 24 months survival of all grafts
Time Frame: Graft survival was monitored from transplant date until retransplantation or death up to 2 years as in SRTR data file October 2015
Population: All grafts transplanted from donors in the RIPNOD trial and in whom recipient records are available in SRTR were included in this analysis. Graft loss is defined as retransplantation or death during the 24 months post-transplant.
Measure: Number; unit: percentage of all grafts
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 523 | 489
percentage of all grafts
  6 months graft survival | 91.3 | 94.6
  12 months | 88.8 | 92.2
  24 months | 82.2 | 87.8
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.03, Log Rank; This is an unadjusted comparison

15. Post Hoc Outcome: Death-Censored Kidney Graft Survival at 6, 12 and 24 Months
Description: kidney graft survival censored for death with functioning graft
Time Frame: Kidney graft survival was monitored from transplant date until retransplantation or death up to 2 years as in SRTR data file October 2015
Population: Included were kidneys transplanted alone or with pancreas. All kidney grafts transplanted from donors in the RIPNOD trial and in whom recipient records are available in SRTR were included in this analysis. Kidney graft loss is defined as loss of functioning graft or retransplantation during the 24 months post-transplant.
Measure: Number; unit: percentage of participants
Groups:
- No RIPC: Kidneys in this group were recovered from donors in the No RIPC arm.
- RIPC: Kidneys in this group were recovered from donors in the RIPC arm.
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 247 | 235
percentage of participants
  Death censored kidney survival: 6 months | 94.2 | 99.1
  12 months | 92.5 | 96.8
  24 months | 87.4 | 96
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.01, Log Rank; Results of adjusted Cox proportional hazard analyses for six month death-censored kidney graft survival are shown below; Cox Proportional Hazard = 0.19, 95% CI 2-sided [0.04 to 0.90] — The proportional hazard ratio favors RIPC group

16. Post Hoc Outcome: Recipient Survival
Description: Kaplan-Meier estimates of 6, 12 and 24 months survival of all recipients
Time Frame: Recipient survival was monitored from transplant date until death up to 2 years as in SRTR data file October 2015
Population: All recipients of organs from donors in the RIPNOD trial and in whom recipient records are available in SRTR were included in this analysis
Measure: Number; unit: percentage of participants
Groups:
- No RIPC: The recipients in this group received one or more organs from donors in the No RIPC arm of the RIPNOD trial.
- RIPC: The recipients in this group received one or more organs from donors in the RIPC arm of the RIPNOD trial
Arm/Group | No RIPC | RIPC
Number analyzed (Participants) | 494 | 458
percentage of participants
  Recipient survival: 6 months | 92 | 94.1
  12 months | 90.0 | 91.5
  24 months | 84.4 | 87.1
Statistical Analysis 1: Comparison: No RIPC vs RIPC; Test type: Superiority or Other; p = 0.37, Log Rank; This is an unadjusted comparison

ADVERSE EVENTS:
Description: Adverse events to be collected were not identified or defined a priori. In donors, data were collected from enrollment to organ recovery; recipient data for DGF in kidney recipients were abstracted from transplantation to last follow up to 2 years in SRTR. Lack of information in SRTR precluded analyses regarding the severity of DGF. Submitted followup data was available at 6, 12 and 24 months in 97.5%, 75.5% and 38.8% of recipients, respectively. Updated SRTR recipient data has been requested.
Groups:
- No RIPC, Kidney Recipients: Recipients in this group received kidneys from donors who did not receive remote ischemic preconditioning (No RIPC group)
- RIPC, Kidney Recipients: Recipients in this group received kidneys from donors who received two RIPC interventions
- No RIPC, All Organ Recipients: Recipients in this group received organs from donors who did not receive remote ischemic preconditioning (No RIPC)
- RIPC, All Organ Recipients: Recipients in this group received organs from donors who received two RIPC interventions
- No RIPC, Donors: Donors in this group did not receive remote ischemic preconditioning (RIPC)
- RIPC, Donors: Donors in this group received two RIPC interventions
Arm/Group | No RIPC, Kidney Recipients | RIPC, Kidney Recipients | No RIPC, All Organ Recipients | RIPC, All Organ Recipients | No RIPC, Donors | RIPC, Donors
Serious Adverse Events (participants affected / at risk) | 45/247 | 51/235 | 81/494 | 54/458 | 8/166 | 14/155
Other Adverse Events (participants affected / at risk) | 0/247 | 0/235 | 0/494 | 0/458 | 0/166 | 0/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | No RIPC, Kidney Recipients (N=247) | RIPC, Kidney Recipients (N=235) | No RIPC, All Organ Recipients (N=494) | RIPC, All Organ Recipients (N=458) | No RIPC, Donors (N=166) | RIPC, Donors (N=155)
DGF in kidney recipients (Renal and urinary disorders) | 45 (45) | 51 (51) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) — DGF defined as dialysis within the first week after kidney transplant
Kidney rejection (Renal and urinary disorders) | 17 (17) | 13 (13) | 0/0 (0) | 0/0 (0) | 0 | 0 — Kidney recipients that had an episode of rejection within the first 6 months
Grafts lost (General disorders) | 26 (26) | 10 (10) | 81 (81) | 52 (52) | 0/0 (0) | 0/0 (0) — Number of grafts lost in all recipients
Recipient Deaths (General disorders) | 23 (23) | 20 (20) | 69 (69) | 54 (54) | 0/0 (0) | 0/0 (0) — Recipient Deaths in all recipients
Number of Donors from which no Organs recovered (General disorders) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 0/0 (0) | 8 (8) | 14 (14)

LIMITATIONS AND CAVEATS:
1) Bias from variation in the intervention between two sites; 2) Lack of blinding; 3) Inadequate data precludes analyses of ejection fraction; 4) Data on some of the other secondary outcomes were not available for all donors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No